CLINICAL TRIAL: NCT00333372
Title: To Evaluate the Efficacy of Z-338 in Subjects With Functional Dyspepsia, Focusing on the Assessment of Subjective Symptoms
Brief Title: To Evaluate the Efficacy of Z-338 in Subjects With Functional Dyspepsia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Zeria Pharmaceutical (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 99010207
Record Dates: First submitted 2006-06-02; First posted 2006-06-05 (Estimated); Last update posted 2009-01-14 (Estimated); Status verified 2009-01

CONDITIONS: Functional Dyspepsia
MeSH Terms: interventions — Z 338

INTERVENTIONS:
Drug: Z-338

SUMMARY:
To Evaluate the efficacy of Z-338 in subjects with Functional Dyspepsia, focusing on the assessment of subjective symptoms in order to further determine the optimal dosage and efficacy parameters for PhaseIII clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Postprandial fullness, upper abdominal bloating and/or early satiety should be at least moderate for 2 days or more at the 7 days at Visit 1
* upper abdominal pain, upper abdominal discomfort, postprandial fullness, upper abdominal bloating, early satiety, nausea, vomit and belching should be at least moderate for at least 2 symptoms for 2 days or more at the 7 days at Visit 1

Exclusion Criteria:

* subjects taht heartburn should be the most bothersome symptom
* Subjects presenting with primary complaints relieved by stool movements (IBS)
* Subjects with diabetes by treatment
* Subjects taht heartburn should be more than moderate

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 440
Dates: Start 2006-04

PRIMARY OUTCOMES:
General impression at last visit

SECONDARY OUTCOMES:
General impression at each week
Individual symptom score

CONTACTS AND LOCATIONS:
Overall Officials: Michio Hongo, Professor, Study Director — Tohoku University Hospital
Locations (1):
- Tohoku University, Sendai, Japan